CLINICAL TRIAL: NCT01104493
Title: A Prospective, Randomized, Double-Blind, Placebo-Controlled Study to Assess the Safety of a New 6:2 Influenza Virus Reassortant
Brief Title: A Clinical Study to Assess the Safety of a New Influenza Vaccine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Robert A. Gasser, Jr., MD, MedImmune LLC
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CD-VA-FluMist-1045
Record Dates: First submitted 2010-04-13; First posted 2010-04-15 (Estimated); Results first posted 2011-07-14 (Estimated); Last update posted 2011-07-18 (Estimated); Status verified 2011-07

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Single dose of monovalent vaccine
  Interventions: Biological: Monovalent Frozen FluMist®
- 2 (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Monovalent Frozen FluMist® — Single dose of monovalent vaccine (240 subjects) by intranasal spray on Study Day 1.
  Arms: 1
Other: Placebo — Single dose of placebo (60 subjects) by intranasal spray on Study Day 1
  Arms: 2

SUMMARY:
To assess the safety of a new influenza virus vaccine containing a new virus strain in healthy patients prior to the release of the vaccine.

DETAILED DESCRIPTION:
This prospective, randomized, double-blind, placebo-controlled release study will enroll approximately 300 healthy adults 18-49 years of age. Eligible subjects will be randomly assigned in a 4:1 fashion to receive a single dose of monovalent vaccine or placebo by intranasal spray. This study will be conducted at multiple sites in the United States. Randomization will be stratified by site.

Each subject will receive one dose of investigational product on Study Day 1. The duration of study participation for each subject is the time from receipt of investigational product through 180 days after receipt of investigational product.

To summarize the primary safety phase data (Study Days 1-8), the study will be unblinded to the analysis team at MedImmune after all data through at least Study Day 8 are locked.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 through 49 years of age (not yet reached their 50th birthday) at the time of investigational product administration
* Healthy by medical history and physical examination
* Written informed consent and any locally required authorization (eg, Health Insurance Portability and Accountability Act in the United States of America, European Union [EU] Data Privacy Directive in the EU) obtained from the subject/legal representative prior to performing any protocol-related procedures, including screening evaluations
* Female subjects of child-bearing potential, (ie, unless at least 2 years postmenopausal, surgically sterile [eg, bilateral tubal ligation, bilateral oophorectomy, or hysterectomy], has sterile male partner, or practices abstinence) must use an effective method of avoiding pregnancy (including oral, transdermal, or implanted contraceptives, intrauterine device, female condom with spermicide, diaphragm with spermicide, cervical cap, or use of a condom with spermicide by the sexual partner) for 30 days prior to administration of investigational product, and must agree to continue using such precautions for 60 days after investigational product administration. In addition, the subject must also have a negative urine or blood pregnancy test at screening and, if screening and Day 1 do not occur on the same day, on the day of vaccination prior to randomization.
* Males, unless surgically sterile must use an effective method of birth control with a female partner and must agree to continue using such contraceptive precautions for at least 30 days after dosing with investigational product (from Study Day 1 through Study Day 31)
* Subject available by telephone
* Ability to understand and comply with the requirements of the protocol, as judged by the investigator
* Ability to complete follow-up period of 180 days after dosing as required by the protocol

Exclusion Criteria:

* History of hypersensitivity to any component of the vaccine, including egg or egg protein or serious, life threatening, or severe reactions to previous influenza vaccinations
* History of hypersensitivity to gentamicin
* Any condition for which the inactivated influenza vaccine is indicated, including chronic disorders of the pulmonary or cardiovascular systems (eg, asthma), chronic metabolic diseases (eg, diabetes mellitus), renal dysfunction, or hemoglobinopathies that required regular medical follow-up or hospitalization during the preceding year Note: A history of asthma that requires regular medical follow-up or hospitalization during the preceding 2 years is exclusionary. Investigator judgment is required to determine whether or not a subject has a history of asthma; however, for adult subjects, a remote history of wheezing or a remote diagnosis of asthma that the investigator does not consider to be relevant to current health does not need to be considered to be a history of asthma. For example, childhood asthma that has not required treatment in adulthood is not necessarily exclusionary
* Acute febrile (> 100.0°F oral or equivalent) and/or clinically significant respiratory illness (eg, cough or sore throat) within 14 days prior to randomization
* Any known immunosuppressive condition or immune deficiency disease, including human immunodeficiency virus (HIV) infection, or ongoing immunosuppressive therapy
* History of Guillain-Barré syndrome
* A household contact who is severely immunocompromised (eg, hematopoietic stem cell transplant recipient, during those periods in which the immunocompromised individual requires care in a protective environment); additionally, subject should avoid close contact with severely immunocompromised individuals for at least 21 days after receipt of investigational product
* Receipt of any investigational agent within 30 days prior to randomization, or expected receipt through 30 days after the dose of investigational product
* Receipt of any non-study vaccine within 30 days prior to randomization, or expected receipt through 30 days after receipt of investigational product
* Expected receipt of antipyretic or analgesic medication on a daily or every other day basis from randomization through 14 days after receipt of investigational product Note: A daily dose of up to 81 mg of aspirin for prophylactic use is not considered a contraindication to enrollment.
* Administration of intranasal medications within 14 days prior to randomization, or expected receipt through 14 days after administration of investigational product
* Receipt of influenza antiviral therapy or antiviral agents within 48 hours prior to investigational product administration or expected receipt of influenza antiviral therapy or antiviral agents through 14 days after receipt of each dose of investigational product
* Known or suspected mitochondrial encephalomyopathy
* Nursing mother
* Any condition (eg, chronic cough) that, in the opinion of the investigator, would interfere with evaluation of the investigational product or interpretation of subject safety or study results
* Employees of the clinical study site, any other individuals involved with the conduct of the study, or immediate family members of such individuals

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2010-05; Primary Completion 2010-06 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert A. Gasser, Jr., M.D., Study Director — MedImmune LLC
Locations (3):
- United States (3):
  - Miami Research Associates, South Miami, Florida
  - Clinical Research Atlanta, Stockbridge, Georgia
  - Columbia Research Group, Inc, Portland, Oregon

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Three investigators at 3 clinical research units in the United States of America (USA) enrolled 300 subjects in May, 2010.
Groups:
- Monovalent Influenza Virus Vaccine: Frozen monovalent vaccine containing the new strain was supplied in intranasal sprayers containing a total volume of 0.2 mL of sucrose phosphate/concentrated gelatin-arginine-glutamate buffer, egg allantoic fluid, and approximately 10^7 fluorescent focus units of influenza virus type A/Perth/16/2009 (H3N2) virus. A single dose of investigational product was administered on Day 1.
- Placebo: Placebo was supplied in intranasal sprayers containing 0.2 mL of sucrose phosphate/concentrated gelatin-arginine-glutamate buffer. A single dose of investigational product was administered on Day 1.
Period: Overall Study
Arm/Group | Monovalent Influenza Virus Vaccine | Placebo
Started | 240 | 60
Completed | 240 | 58
Not Completed | 0 | 2
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Monovalent Influenza Virus Vaccine | Placebo | Total
Number analyzed (Participants) | 240 | 60 | 300
Age Continuous [Mean (Standard Deviation); unit: years] | 32.5 (8.8) | 32.4 (8.3) | 32.5 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 127 | 29 | 156
  Male | 113 | 31 | 144

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Reporting Fever, Defined as Oral Temperature ≥ 101°F
Description: A comparison of the rate of fever (oral temperature ≥ 101°F) reported during the 7 days post administration of investigational product between the monovalent vaccine and placebo groups.
Time Frame: Study Days 1-8
Population: All subjects who received a single dose of investigational product (monovalent vaccine = 240; placebo = 60)
Measure: Number; unit: Percentage of participants
Arm/Group | Monovalent Influenza Virus Vaccine | Placebo
Number analyzed (Participants) | 240 | 60
Percentage of participants | 0.4 | 0.0
Statistical Analysis 1: Comparison: Monovalent Influenza Virus Vaccine vs Placebo; Comparison of the rate of fever between the 2 treatment groups was based on the upper limit of the two-sided 95% exact confidence intervals (CIs) for the rate increase (Monovalent vaccine minus Placebo) evaluated against the prespecified equivalence criterion of 5 percentage points; Test type: Non-Inferiority or Equivalence — H0 (null): Rate difference ≥ 5 percentage points This corresponded to a null hypothesis of: HA (alternative): rate difference < 5 percentage points; score statistic; rate difference = 0.4, 95% CI 2-sided [-5.2 to 2.6]

2. Secondary Outcome: Percentage of Participants Reporting Any Solicited Symptom
Description: Solicited symptoms were events that were considered likely to occur post dosing. Solicited symptoms for this study are listed below.
Time Frame: Study Days 1-8
Population: All subjects who received a single dose of investigational product (monovalent vaccine = 240; placebo = 60)
Measure: Number; unit: Percentage of participants
Arm/Group | Monovalent Influenza Virus Vaccine | Placebo
Number analyzed (Participants) | 240 | 60
Percentage of participants
  Any symptom | 33.8 | 40.0
  Fever > 100F | 0.8 | 0.0
  Fever > 102F | 0.0 | 0.0
  Fever > 103F | 0.0 | 0.0
  Runny nose | 13.3 | 18.3
  Sore throat | 8.8 | 5.0
  Cough | 7.5 | 6.7
  Vomiting | 0.8 | 0.0
  Muscle aches | 5.8 | 3.3
  Chills | 2.5 | 1.7
  Decreased activity (tiredness) | 8.3 | 6.7
  Headache | 16.7 | 16.7

3. Secondary Outcome: Percentage of Participants Reporting Any Adverse Event.
Description: An adverse event (AE) was defined as: Any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Time Frame: Study Days 1-8
Population: All subjects who received a single dose of investigational product (monovalent vaccine = 240; placebo = 60)
Measure: Number; unit: Percentage of participants
Arm/Group | Monovalent Influenza Virus Vaccine | Placebo
Number analyzed (Participants) | 240 | 60
Percentage of participants | 3.8 | 3.3

4. Secondary Outcome: Percentage of Participants Reporting Any Solicited Symptom.
Description: as for outcome 2
Time Frame: Study Days 1-15
Population: All subjects who received a single dose of investigational product (monovalent vaccine = 240; placebo = 60)
Measure: Number; unit: Percentage of participants
Arm/Group | Monovalent Influenza Virus Vaccine | Placebo
Number analyzed (Participants) | 240 | 60
Percentage of participants
  Any Symptom | 38.3 | 50.0
  Fever > 100F | 1.7 | 1.7
  Fever ≥ 101F | 0.8 | 1.7
  Fever > 102F | 0.0 | 0.0
  Fever > 103F | 0.0 | 0.0
  Runny nose | 17.1 | 21.7
  Sore throat | 10.8 | 8.3
  Cough | 8.8 | 6.7
  Vomiting | 1.3 | 0.0
  Muscle aches | 7.5 | 6.7
  Chills | 3.3 | 1.7
  Decreased activity (tiredness) | 8.8 | 8.3
  Headache | 19.2 | 25.0

5. Secondary Outcome: Percentage of Participants Reporting Any Adverse Event.
Description: as for outcome 3
Time Frame: Study Days 1-15
Population: All subjects who received a single dose of investigational product (monovalent vaccine = 240; placebo = 60)
Measure: Number; unit: Percentage of participants
Arm/Group | Monovalent Influenza Virus Vaccine | Placebo
Number analyzed (Participants) | 240 | 60
Percentage of participants | 4.2 | 3.3

6. Secondary Outcome: Percentage of Participants Reporting at Least One Serious Adverse Event (SAE) or New Onset Chronic Disease (NOCD), Study Days 1-29
Description: SAEs were those that resulted in death; were life-threatening; resulted in inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability or incapacity; were a congenital anomaly/birth defect in the offspring of a study participant; or were a medical event that may have jeopardized the subject and may have required medical or surgical intervention to prevent one of the outcomes listed above. An NOCD was a newly diagnosed medical condition of a chronic, ongoing nature and assessed by the investigator as medically significant.
Time Frame: Study Days 1-29
Population: All subjects who received a single dose of investigational product (monovalent vaccine = 240; placebo = 60)
Measure: Number; unit: Percentage of participants
Arm/Group | Monovalent Influenza Virus Vaccine | Placebo
Number analyzed (Participants) | 240 | 60
Percentage of participants
  Total participants reporting ≥ one SAE | 0.0 | 0.0
  Total participants reporting ≥ one NOCD | 0.0 | 0.0

7. Secondary Outcome: Percentage of Participants Reporting at Least One Serious Adverse Event (SAE) or New Onset Chronic Disease (NOCD), Study Days 1-181
Description: as for outcome 6
Time Frame: Study Days 1-181
Population: All subjects who received a single dose of investigational product (monovalent vaccine = 240; placebo = 60)
Measure: Number; unit: Percentage of participants
Arm/Group | Monovalent Influenza Virus Vaccine | Placebo
Number analyzed (Participants) | 240 | 60
Percentage of participants
  Total participants reporting ≥ one SAE | 1.3 | 0.0
  Total participants reporting ≥ one NOCD | 0.0 | 0.0

ADVERSE EVENTS:
Time Frame: From the time that written informed consent was obtained, adverse events were collected through Study Day 15 after receipt of investigational product and serious adverse events were collected through Study Day 181 after receipt of investigational product.
Arm/Group | Monovalent Influenza Virus Vaccine | Placebo
Serious Adverse Events (participants affected / at risk) | 3/240 | 0/60
Other Adverse Events (participants affected / at risk) | 6/240 | 2/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Monovalent Influenza Virus Vaccine (N=240) | Placebo (N=60)
oesophageal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
menometrorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Monovalent Influenza Virus Vaccine (N=240) | Placebo (N=60)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (2)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Depressed mood (Psychiatric disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.